CLINICAL TRIAL: NCT00980603
Title: A Randomized Phase II Study of Docetaxel vs. Docetaxel Plus Cisplatin vs. Docetaxel Plus S-1 as Second-line Chemotherapy After Cisplatin Plus S-1 or Capecitabine in Metastatic Gastric Cancer
Brief Title: Docetaxel Versus Docetaxel Plus Cisplatin Versus Docetaxel Plus S-1 as Second-line Chemotherapy in Metastatic Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Seoul National University Bundang Hospital (Other); Chungbuk National University Hospital (Other); Gachon University Gil Medical Center (Other)
Responsible Party: Sook Ryun Park/Dr., Research Institute and Hospital, National Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-07-296
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; metastatic; docetaxel; cisplatin; S-1
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — Docetaxel; Cisplatin; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- docetaxel (Active Comparator)
  Interventions: Drug: docetaxel
- doctaxel plus cisplatin (Experimental)
  Interventions: Drug: docetaxel, cisplatin
- docetaxel plus S-1 (Experimental)
  Interventions: Drug: docetaxel, S-1

INTERVENTIONS:
Drug: docetaxel — docetaxel 75 mg/m2, IV on day 1 of each 3 week cycle until progression or unacceptable toxicity develops
  Arms: docetaxel
Drug: docetaxel, cisplatin — docetaxel 60 mg/m2 and cisplatin 60 mg/m2, IV on day 1 of each 3 week cycle until progression or unacceptable toxicity develops
  Arms: doctaxel plus cisplatin
Drug: docetaxel, S-1 — docetaxel 60 mg/m2 IV on day 1 and S-1 30 mg/m2 bid PO on days 1-14 of each 3 week cycle until progression or unacceptable toxicity develops
  Arms: docetaxel plus S-1

SUMMARY:
The purpose of this study is to assess efficacy and safety of docetaxel alone, docetaxel plus cisplatin, and docetaxel plus S-1 in patients with metastatic gastric cancer after failing 1st line chemotherapy with cisplatin plus S-1 or capecitabine

DETAILED DESCRIPTION:
To date, the most commonly used first-line chemotherapies have been based on fluorouracil and/or cisplatin in patients with metastatic gastric cancer. Unfortunately, considerable proportions of patients with metastatic gastric cancer do not respond to first-line chemotherapy and most of the patients who do respond eventually experience disease progression. In the second-line treatment, however, standard therapies are less clearly defined.

Meanwhile, regarding re-challenge of previous failed drugs as a combination with an other newly introduced chemotherapeutic agent, there are few data. Increased expression and activity of thymidylate synthase, which is inhibited by fluoropyrimidine, is regarded to be the main reason for the development of clinical resistance to fluoropyrimidine. Since the cotreatment of docetaxel and 5-fluorouracil decreases the activity and expression of thymidylate synthase and dihydropyrimidine dehydrogenase (5-fluorouracil degradation enzyme), and increases the expression of orotate phosphoribosyl transferase, the addition of docetaxel into S-1 may recover the sensitivity to S-1 in patients previously resistant to S-1.

Several reports found that MDR-1 and MRP-1 are related to cisplatin-resistance; cisplatin induces the overexpression of MRP-1, which reduces intracellular cisplatin accumulation. Since docetaxel suppresses the cisplatin-induced MRP-1 upregulation, the addition of docetaxel into cisplatin may recover the sensitivity to cisplatin in patients previously resistant to cisplatin.

Based on these synergism mechanisms, we speculate that the cotreatment of docetaxel and cisplatin or S-1 has better anti-tumor activity than docetaxel alone in patients resistant to cisplatin or S-1.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed gastric adenocarcinoma with metastatic disease
* Age ≥18 years
* Eastern Cooperative Oncology Group performance status 0-2
* At least one measurable lesion as defined by RECIST
* Only one prior chemotherapy containing both S-1 or capecitabine and cisplatin for metastatic gastric cancer with documented progression of disease occurring during chemotherapy or within 6 months of completion of chemotherapy
* Adequate major organ function:

ANC ≥1,500/mm3, Platelet ≥100,000/mm3, serum bilirubin ≤1.5 x upper limit of normal (ULN), AST/ALT ≤2.5 x ULN (≤5 x ULN if liver metastases are present), creatinine clearance ≥50 ml/min using the calculation formula or 24 hours urine collection

* Patients should sign a written informed consent before study entry

Exclusion Criteria:

* Prior taxane treatment
* Major surgery or radiotherapy less than 4 weeks prior to entry
* NCI CTCAE (version 3.0) adverse events ≥grade 2 except alopecia, fatigue, and weight loss
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome, or inability to take oral medication
* Patients with active gastrointestinal bleeding
* Inadequate cardiovascular function
* Serious concurrent infection or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy
* Other malignancy within the past 3 years except adequately treated non-melanomatous skin cancer, carcinoma in situ of the cervix, or in situ of prostate cancer Gleason≤7
* Psychiatric disorder that would preclude compliance
* Patients receiving a concomitant treatment with drugs interacting with S-1 such as flucytosine, phenytoin, or allopurinol
* Female patients who are pregnant or breast feeding or adults of reproductive potential not employing effective method of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-11 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
response rate | every 2 cycles

SECONDARY OUTCOMES:
time to progression | every 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Sook Ryun Park, Dr., Principal Investigator — Research Institute and Hospital, National Cancer Center Korea
Locations (4):
- South Korea (4):
  - Research Institute and Hospital, National Cancer Center Korea, Goyang
  - Gachon University Gil Hospital, Inchon
  - Chungbuk National University Hospital, Jeonju
  - Seoul National University Bundang Hospital, Seongnam